CLINICAL TRIAL: NCT03033992
Title: Feasibility Trial of Optune for Children With Recurrent or Progressive Supratentorial High-Grade Glioma or Ependymoma, and Feasibility and Efficacy Trial of Optune in Conjunction With Radiation Therapy for Children With Newly Diagnosed DIPG
Brief Title: Optune for Children With High-Grade Glioma or Ependymoma, and Optune With Radiation Therapy for Children With DIPG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NovoCure Ltd. (Industry); American Lebanese Syrian Associated Charities (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-048; UM1CA081457 (NIH); NCI-2016-00926 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-048 (Other: Pediatric Brain Tumor Consortium); PBTC-048 (Other: CTEP)
Record Dates: First submitted 2017-01-17; First posted 2017-01-27 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Malignant Glioma; Ependymoma; Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Glioma; Ependymoma; Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Intervention Model Description: The study includes two independent strata. Stratum 1 is a single-arm safety and feasibility study. While stratum 2 is a phase I/II study which consists of two parts: a phase I component to evaluate the safety and tolerability of concurrent Optune and RT, and a phase II component to evaluate the feasibility of concurrent Optune and RT and the efficacy associated with this approach compared to historical controls.
Masking Description: Open-label single-arm study within each stratum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Optune System) (Experimental): Patients must have a histologically confirmed diagnosis of supratentorial high-grade glioma or supratentorial ependymoma that is recurrent, progressive or refractory. All patients will use the study device Optune System (Tumor Treating Fields, TTFields).
  Interventions: Device: Optune System (NovoTTF-200A System, Tumor Treating Fields, TTFields)
- Treatment (Concurrent Optune/focal radiation therapy followed by Optune-only therapy) (Experimental): Patients must have newly diagnosed DIPG (a typical DIPG on MR imaging, defined as a tumor with a pontine epicenter and diffuse involvement of more than 2/3 of the pons, without histologic confirmation; atypical DIPG undergoing a biopsy and the tumor is a diffuse glioma WHO Grade II-IV with OR without H3 K27M mutation; or pontine lesions that do not meet these MR imaging criteria with histologically confirmed diffuse glioma WHO Grade II-IV with H3 K27M- mutation). This arm will consist of two parts: a phase I component to evaluate the safety and tolerability of concurrent Optune and RT, and a phase II component to evaluate the feasibility of concurrent Optune and RT and the efficacy associated with this approach compared to historical controls.
  Interventions: Combination Product: Concurrent Optune and RT followed by Optune System alone

INTERVENTIONS:
Device: Optune System (NovoTTF-200A System, Tumor Treating Fields, TTFields) — The Optune, a.k.a. Tumor Treating Fields (TTFields), will be worn for a minimum of 18 hours a day, with a recommendation of 22 hours/day for at least 23 days in a 28-day cycle. Cycle 1 includes 7 days training period, followed by 28 days treatment (total 35 days). The patients will receive multiple 28-day cycles of continuous Optune treatment. In the absence of treatment related serious adverse events or disease progression, Optune will continue up to 26 cycles.
  Other Names: Optune System (NovoTTF-200A System)
  Arms: Treatment (Optune System)
Combination Product: Concurrent Optune and RT followed by Optune System alone — In Stratum II patients will be treated with standard of care focal RT concurrently with Optune followed by Optune treatment. This study specifies a 1 cm clinical target volume margin.The duration of the first cycle of therapy will be from Day 1 of RT to 14 days after completion of RT (approximately 8 weeks total). Subsequent cycles of therapy will be 28 days in duration. The Optune device will be worn for a minimum of 18 hours/day, with a recommendation of 22 hours/day. For the phase I part, the initial treatment will involve RT delivery with Optune arrays remaining in place but turned off. If this is not tolerated, two treatment de-escalation levels are planned, Specifically, Level -1: remove the Optune arrays during RT delivery and reapply daily after RT; Level -2: initiate Optune therapy after completion of RT. The established safe treatment approach from phase I will be investigated for feasibility and efficacy in phase II. Treatment with Optune may continue for up to 5 years.
  Arms: Treatment (Concurrent Optune/focal radiation therapy followed by Optune-only therapy)

SUMMARY:
This is a multicenter trial of the Optune device to examine the feasibility and to describe the device-related toxicity in children with supratentorial high grade glioma (HGG) or ependymoma (Stratum 1) and to examine the feasibility and efficacy of concurrent Optune and standard focal radiation therapy (RT) in children with newly diagnosed diffuse intrinsic pontine glioma (DIPG) (Stratum 2).

DETAILED DESCRIPTION:
The primary objectives of Stratum 1 are: 1) to evaluate the feasibility of treatment with Optune in pediatric patients with recurrent/refractory/progressive supratentorial malignant glioma or ependymoma, and 2) to describe the Optune device treatment-related toxicities in children with recurrent/refractory/progressive supratentorial malignant glioma or ependymoma.

The primary objectives of Stratum 2 are: 1) to describe the safety and tolerability of concurrent Optune therapy and RT (Phase I component), 2) to evaluate the feasibility of treatment with concurrent Optune and RT (Phase II component), and 3) to estimate the overall survival (Phase II component) in children and adolescents with newly diagnosed DIPG treated with concurrent Optune therapy and standard RT.

The Optune System produces alternating electrical fields, called tumor treatment fields (TTFields) by means of 4 transducer arrays placed on the shaved scalp. The very low intensity, intermediate frequency electric fields impair the growth of tumor cells through the arrest of cell division and inducing apoptosis. Preclinical studies have demonstrated TTFields synergistically enhance the efficacy of irradiation in glioma cell lines.

Optune will be worn for a minimum of 18 hours a day, with a recommendation of 22 hours/day for at least 23 days in a 28-day cycle. Treatment may continue up to 26 cycles in Stratum 1 and Optune treatment may continue for up to 5 years in Stratum 2 if the participant is deriving benefit and in the absence of significant treatment-related toxicity. Patients will be followed for 2 years from the cessation of protocol treatment in Stratum 1, and for 3 years from the cessation of Optune device treatment in Stratum 2 for the monitoring of unexpected later developing toxicities and to document disease progression, event-free and overall survival.

For patients in Stratum 1, the therapy will be deemed feasible for patients who are able to use the device for ≥ 18 hours/day for at least 23 days out of 28 days of cycle one (feasibility assessment period). A total of 20 patients need to be assessed with an interim analysis to be conducted after the first 11 patients. Kaplan-Meier estimates of EFS for all eligible patients who use the device for at least 1 day will be provided separately for the two histology-based cohorts i.e. HGG and Ependymoma.

For patients in Stratum 2, the study will consist of two parts: a phase I portion to evaluate the safety and tolerability of concurrent Optune and RT; and a phase II portion to evaluate the feasibility and efficacy of concurrent Optune and standard RT. The therapy will be deemed feasible for patients who are able to use the device for ≥ 18 hours/day for at least 40 of the 49 days of the feasibility assessment period of cycle one, which consists of concurrent Optune and RT. Up to 18 evaluable patients may need to be assessed for the phase I component. A total of 30 patients need to be assessed for the phase II component (6 of whom will be counted from the phase I component). The design also incorporates 2 interim analyses for futility assessed when 9 and 14 events are observed.

ELIGIBILITY:
Inclusion Criteria:

* Age: at the time of enrollment Stratum 1: ≥ 5 years but ≤ 21 Stratum 2: ≥ 3 years but ≤ 21
* Diagnosis:

Stratum 1: Patients must have a histologically confirmed diagnosis of supratentorial high-grade glioma or supratentorial ependymoma that is recurrent, progressive or refractory.

Stratum 2: Patients with newly diagnosed DIPG

* Patients with a typical DIPG on MR imaging, defined as a tumor with a pontine epicenter and diffuse involvement of more than 2/3 of the pons, are eligible without histologic confirmation.
* Note: Patients with typical DIPG who undergo a biopsy are eligible provided the tumor is a diffuse glioma WHO Grade II-IV with OR without H3 K27M mutation.
* Patients with pontine lesions that do not meet these MR imaging criteria will be eligible if there is histologic confirmation diffuse glioma WHO Grade II-IV with H3 K27M-mutation.

  * Disease Status: Patients must have bi-dimensionally measurable disease, defined as at least one lesion that can be accurately measured in at least two planes

Stratum 1:

* This disease must be located primarily in the supratentorial region
* Patients with significant disease that is metastatic outside of the supratentorial region are ineligible

Stratum 2:

* This disease must be located primarily in the pons

  * Prior Therapy:

Stratum 1: Patients must have recovered from the acute treatment related toxicities (defined as ≤ grade 1) of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

Stratum 2: Patients may not have had any prior antitumor therapy except surgery and/or steroids.

• Myelosuppressive Chemotherapy: Patients must have received last dose of known myelosuppressive chemotherapy >21 days prior to enrollment; >42 days if nitrosourea.

* Biologic Agent: Biologic agent must have recovered from any acute toxicity potentially related to the agent and received their last dose of the biologic agent > 7 days prior to study enrollment.

  - For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
* Immunomodulatory treatment: Patient must have received the last dose >21 days prior to enrollment.

  - Monoclonal antibody treatment and agents with known prolonged half-lives: Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 28 days prior to study enrollment. Radiation:
  * Stratum 1: Patients must have had their last fraction of:

    - Craniospinal irradiation (>24Gy) or total body irradiation or radiation to ≥ 50% of pelvis ≥ 42 days prior to enrollment
    * Focal irradiation ≥ 14 days prior to enrollment
    * Local palliative irradiation (small port) ≥ 14 days
  * Stratum 2: Patients must not have received any radiotherapy prior to enrollment. If clinically indicated, enrolled patients may receive up to 5 fractions of radiotherapy prior to starting Optune therapy.
* Surgery:

  o Stratum 1: Optune device application start date must be at least 4 weeks (28 days) from CNS surgical procedure. Excluding VP shunts, Endoscopic Third Ventriculostomy (ETV) for which treatment could start 10 days post procedure. Non-CNS surgical procedures such as but not limited to central venous catheter insertion at the discretion of treating physician and study chair.

  o Stratum 2: Radiation therapy and Optune device application start date must be at least 5 days after the date of a tumor biopsy if obtained.
* Inclusion of Women and Minorities: Both males and females of all races and ethnic groups are eligible for this study.
* Neurologic Status:

  * Stratum 1: Patients with neurological deficits should be stable for a minimum of 1 week prior to enrollment.
  * Stratum 2: Stable neurologic deficits are not an eligibility criterion for Stratum 2.

Performance Status: Stratum 1: Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) assessed within two weeks of enrollment must be ≥ 60. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score. There are no performance status requirements for Stratum 2 patients.

• Organ Function: Stratum 1 patients must have organ and marrow function as defined below: Absolute neutrophil count ≥ 1.0 X 109/L; Platelets ≥ 100 X 109/L (transfusion independent); Hemoglobin ≥8g/dl (may receive transfusions); Total bilirubin ≤1.5 times institutional upper limit of normal (ULN); ALT(SGPT) ≤3 times institutional upper limit of normal; AST(SGOT) ≤3 times institutional upper limit of normal; Albumin ≥2 g/dl. Serum creatinine based on age/gender as noted below. Patients that do not meet the criteria below but have a 24 hour Creatinine Clearance or GFR (radioisotope or iothalamate) ≥ 70 ml/min/1.73 m2 are eligible.

Age Maximum Serum Creatinine (mg/dL) 3 to < 6 years 0.8 (Male) 0.8 (Female); 6 to < 10 years 1 (Male) 1 (Female); 10 to < 13 years 1.2 (Male) 1.2 (Female); 13 to < 16 years 1.5 (Male) 1.4 (Female);

* 16 years 1.7 (Male) 1.4 (Female).

  * Stratum 2: Patients must have adequate organ and marrow function as defined below:

    o Absolute neutrophil count ≥ 1.0 X 109/L

    o Platelets ≥ 100 X 109/L (transfusion independent)

    o Hemoglobin ≥8g/dl (may receive transfusions)
  * Head circumference: Patients must have minimum head circumference of 44 cm.
  * Compliance in Optune Device Usage:

    * Stratum 1: Patients must be willing to use the Optune device ≥18 hours/day for at least 23 days in a 28-day cycle, and keep head shaved throughout treatment.
    * Stratum 2: During concurrent Optune therapy and RT, patients must be willing to use the Optune device ≥18 hours/day for at least 40 of the 49 days of the duration of the feasibility period. During subsequent cycles of Optune therapy alone, patients must be willing to use the Optune device ≥18 hours/day for at least 23 days in a 28-day cycle. During concurrent Optune therapy and RT and Optune therapy alone, patients must be willing to keep their head shaved throughout treatment.
  * Pregnancy Status: Female patients of childbearing potential must have a negative serum or urine pregnancy test.
  * Pregnancy Prevention: Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.
  * Informed Consent: The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document according to institutional guidelines.
  * Steroids:

    o Stratum 1: If patient is on corticosteroids, the dose must be stable or decreasing for at least 5 days prior to enrollment.
    * Stratum 2: There are no eligibility requirements for corticosteroid dosing for Stratum 2.

Exclusion Criteria:

* Systemic Illness: Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results.
* Other Malignancy: Patients with a history of any other malignancy.
* Concurrent Therapy: Patients who are receiving any other anticancer or investigational drug therapy are not eligible.
* Inability to Participate: Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to device usage plan, other study procedures, and study restrictions.
* Stratum 1 Tumor Location: Patients with primarily infra-tentorial or spinal cord tumor are not eligible.
* Tumor Dissemination: Patients for who clinical suspicion is present of metastatic disease in the CSF or Spine must have MRI of Spine and CSF obtained (Lumbar puncture or through ommaya, EVD or Shunt) with negative cytology. Patients with CSF that is positive for tumor cells or metastatic disease found on MRI are ineligible.
* Skull Defects: Patients with major skull defects (such as missing bone without replacement) are not eligible.
* Neurological Disorder: Patients with active implanted electronic devices in the brain or spinal cord such as programmable VP shunts, deep brain stimulators, vagus nerve stimulators, are not eligible.
* Cardiac Disorder: Patients with pacemaker, defibrillator, or documented significant arrhythmia, are not allowed.
* Intracranial Objects: Patients with foreign body intracranially, such as bullet fragments, are not allowed, with the exception of VP-shunts (non-programmable) and Ommaya catheters.
* Allergy: Patients with history of hypersensitivity to conductive hydrogel are not eligible.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2031-05-22 (Estimated); Study Completion 2031-07-21 (Estimated)

PRIMARY OUTCOMES:
The feasibility of treatment with the Optune device in pediatric patients with recurrent/refractory/progressive supratentorial malignant glioma and ependymoma. | days 8 through 35 of cycle 1
  Stratum 1: Device Usage Compliance will be reported to assess the feasibility of the device treatment.
The Optune device treatment-related toxicities in children with recurrent/refractory/progressive supratentorial malignant glioma and ependymoma. | 2 years
  Stratum 1: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0.
The type and frequency of Device Limiting Toxicities (DLTs) associated with the Optune treatment given concurrently with RT in children and adolescents with newly diagnosed DIPG. | 5 years
  Stratum 2:The number of participants with DLTs per protocol Section 5.4.
The feasibility of concurrent Optune therapy and RT in children and adolescents with newly diagnosed DIPG. | days 8 through 56 of cycle 1 (days 8 through 35 of cycle 1 if the second dose de-escalation is utilized for phase II)
  Stratum 2: Device Usage Compliance will be reported to assess the feasibility of the device treatment when administered concurrent with RT. The device treatment will be considered feasible for a patient who use the device for ≥18 hours/day for at least 40 of 49 days (23 of 28 days if the second dose de-escalation is utilized for phase II) of the feasibility period of Cycle 1.
The overall survival | 3 years
  Stratum 2: OS is defined as time from enrollment to death due to any cause.

SECONDARY OUTCOMES:
The Response Rate | 2 years
  Stratum 1: The response rate is calculated according to the bi-dimensional tumor measurement at the end of treatment compared with the baseline measurements.
The Event-Free Survival | 2 years
  Stratum 1: The event-free survival is the interval of time between date of initiation of protocol treatment and minimum date of documentation of progressive disease, second malignancy, death due to any cause, or date of last follow-up.
The association of anti-tumor activity with compliance in Optune device use within the context of a small feasibility study. | 2 years
  Stratum 1:The anti-tumor activity will be classified as complete response, partial response, stable disease, and progressive disease per protocol specified criteria. The compliance in Optune device use will be calculated as the actual hours of Optune device usage per day.
The association between the Optune device usage and the health-related quality of life of children and families undergoing this therapy. | 2 years
  Stratum 1:The Quality of Life Scores will be reported at baseline, and with each cycle using PROMIS and Neuro-QoL Stigma, in which the mean score of the general population is 50 and standard deviation is 10.
The association of apparent diffusion coefficient (ADC) values within the tumor and correlate with response to Optune treatment and EFS. | 2 years
  Stratum 1: We will summarize the tumor-type specific ADC value at baseline and at various times on treatment as well as within-patient changes over time. The ADC value of responders will be compared to the ADC value of those with progressive diseases at baseline and over time.
The Response Rate | 3 years
  Stratum 2: The response rate is calculated according to the bi-dimensional tumor measurement at the end of treatment compared with the baseline measurements.
The Event-Free Survival | 3 years
  Stratum 2: The event-free survival will be measured from the date of initial treatment to the earliest date of disease progression, second malignancy or death for any reason for patients who fail; and to the date of last contact for patients who remain at risk for failure.
Compliance rate | 3 years
  Stratum 2: A patient will be considered compliant if he/she uses the device for ≥18 hours/day for at least 23 days in a 28-day cycle.
The Quality of Life Scores | 3 years
  The Quality of Life (QoL) Scores will be reported at baseline, and with each cycle using Patient Reported Outcomes Measurement Information System (PROMIS) and Quality of Life in Neurological Disorders (Neuro-QoL) Stigma Scale, in which the mean score of the general population is 50 and standard deviation is 10.
  The PROMIS is rated 0-4 with 0 being "never" (better outcome) and 4 being "almost always," (worse outcome).
  Neuro-QOL Scale is rated 1-5 with 1 being "never" (better outcome) and 5 being "always," (worse outcome).
The association of apparent diffusion coefficient (ADC) values in the tumor with response rate and EFS. | 3 years
  We will summarize the tumor-type specific ADC value at baseline and at various times on treatment as well as within-patient changes over time. The ADC value of responders will be compared to the ADC value of those with progressive diseases at baseline and over time.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Goldman, MD, Principal Investigator — Phoenix Children's Hospital
Locations (11):
- United States (11):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Pediatric Brain Tumor Consortium (PBTC) ensures that high dimensional molecular data generated from PBTC samples will be submitted to the NIH Database of Genotypes and Phenotypes (dbGaP) or other NIH-designated data repository. PBTC is required to make data available to other investigators for use in research projects. An investigator requesting data from published PBTC studies will submit a proposal describing the studies from which data are requested, the requested data, and a list of investigators in the project and their affiliated institutions, along with the investigator's CV to the PBTC Steering Committee for review. Once approved, the requesting investigator will be asked to complete a Data Transfer Agreement before the release of deidentified data. Requests for data are typically only considered once the primary study manuscript has been published though exceptions may be made in the event of long delays in the primary study data publication.
Supporting Information: Study Protocol, ICF, CSR